CLINICAL TRIAL: NCT04956094
Title: Association of Elevated Serum Gamma Glutamyl Transferase (GGT) and Uric Acid at 9-14 Weeks Gestation With the Development of Gestational Diabetes Mellitus (GDM)
Brief Title: GGT and Uric Acid to Predict Gestational Diabetes Mellitus
Acronym: GGTUAGDM
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left the institution.
Sponsor: Mount Carmel Health System (Other)
Collaborators: Mount Carmel Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 210412-1
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-11

CONDITIONS: Gestational Diabetes
Keywords: Pregnancy; Screening; Gamma Glutamyl Transferase; Serum Uric Acid; Sensitivity; Specificity; Predictive Value
MeSH Terms: conditions — Diabetes, Gestational; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- First Trimester Prenatal Visit: Women attending an initial first trimester prenatal visit who will be undergoing a standard blood draw.
  Interventions: Diagnostic Test: GGT/Uric Acid

INTERVENTIONS:
Diagnostic Test: GGT/Uric Acid — Standard laboratory blood testing for GGT and uric acid levels.

SUMMARY:
Gestational Diabetes Mellitus (GDM) is a common metabolic complication of pregnancy defined as new onset hyperglycemia during gestation. GDM conveys significant risk of morbidity and mortality for both mother and infant. An estimated 268,900 infants were born to mothers with GDM in the USA, accounting for approximately 6.9% of births. Although individual correlations have been found between elevated GGT and uric acid levels and later development of GDM, no research has established and validated combined criteria for GGT and uric acid levels that would lead to their use in identifying women at high risk of GDM in the first trimester.

Central Hypothesis: Serum GGT and serum uric acid collected between >9-14.0 weeks gestation will be significantly elevated in women who later develop GDM compared to those who do not. Combined analysis of serum uric acid and GGT levels within the first trimester allows for accurate prediction of the development of GDM.

Study population includes women between 9-14 weeks gestation undergoing a standard first trimester blood draw. Additional blood will be drawn during the standard blood draw to assess GGT and uric acid levels. Research participants will be tracked afterwards to determine whether they tested positive for gestational diabetes during the standard testing process which typically occurs at 24-28 weeks gestation. The data will then be analyzed to estimate the sensitivity, specificity, positive and negative predictive values of the first trimester GGT and uric acid tests. The GGT and uric acid levels which maximize the area under the receiver-operator characteristic curve will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between > 9 weeks and < 14.0 weeks gestation

Exclusion Criteria:

* Known history of or current diagnosis of type I or type II diabetes mellitus
* Known liver disease
* Known kidney disease
* Known history of or current diagnosis of gout
* Known history of alcoholism or current alcohol use
* Multiple gestation
* < 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Females
Study Population: Pregnant women between > 9 weeks and < 14 and 0 weeks gestation presenting to the OB clinic for prenatal care
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients diagnosed with gestational diabetes mellitus | 24-28 weeks
  Diagnosis of gestational diabetes mellitus (GDM) via oral glucose tolerance testing (Carpenter and Coustan criteria)

CONTACTS AND LOCATIONS:
Overall Officials: James Dombroski, MD, Study Chair — Mount Carmel Health System
Locations (1):
- Mount Carmel Health System, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with others. Study data may be requested from the sponsor or investigator.